CLINICAL TRIAL: NCT01463696
Title: A Phase I Study to Evaluate the Safety and Tolerability and Pharmacokinetic/Pharmacodynamics of MK-8242 in Patients With Advanced Solid Tumors
Brief Title: Study of Safety and Pharmacokinetics of MK-8242 in Participants With Advanced Solid Tumors (P07650)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P07650; 2011-001346-15 (EudraCT Number); MK-8242-006 (Other: Merck Protocol Number)
Record Dates: First submitted 2011-10-28; First posted 2011-11-02 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- MK-8242 60 mg BID (Experimental): In Cycle 1, participants received MK-8242 60 mg administered orally (PO) twice a day (BID) on Days 1-6 and PO once daily (QD) in the morning on Day 7 of the 21-day cycle to accommodate pharmacokinetic (PK) sampling. In Cycle 2 and subsequent cycles, participants received MK-8242 60 mg PO BID on Days 1-7 of each 21-day cycle.
  Interventions: Drug: MK-8242
- MK-8242 120 mg BID (Experimental): In Cycle 1, participants received MK-8242 120 mg administered PO BID on Days 1-6 and PO QD in the morning on Day 7 of the 21-day cycle to accommodate PK sampling. In Cycle 2 and subsequent cycles, participants received MK-8242 120 mg PO BID on Days 1-7 of each 21-day cycle.
  Interventions: Drug: MK-8242
- MK-8242 170 mg BID (Experimental): In Cycle 1, participants received MK-8242 170 mg administered PO BID on Days 1-6 and PO QD in the morning on Day 7 of the 21-day cycle to accommodate PK sampling. In Cycle 2 and subsequent cycles, participants received MK-8242 170 mg PO BID on Days 1-7 of each 21-day cycle.
  Interventions: Drug: MK-8242
- MK-8242 250 mg BID (Experimental): In Cycle 1, participants received MK-8242 250 mg administered PO BID on Days 1-6 and PO QD in the morning on Day 7 of the 21-day cycle to accommodate PK sampling. In Cycle 2 and subsequent cycles, participants received MK-8242 250 mg PO BID on Days 1-7 of each 21-day cycle.
  Interventions: Drug: MK-8242
- MK-8242 300 mg BID (Experimental): In Cycle 1, participants received MK-8242 300 mg administered PO BID on Days 1-6 and PO QD in the morning on Day 7 of the 21-day cycle to accommodate PK sampling. In Cycle 2 and subsequent cycles, participants received MK-8242 300 mg PO BID on Days 1-7 of each 21-day cycle.
  Interventions: Drug: MK-8242
- MK-8242 350 mg BID (Experimental): In Cycle 1, participants received MK-8242 350 mg administered PO BID on Days 1-6 and PO QD in the morning on Day 7 of the 21-day cycle to accommodate PK sampling. In Cycle 2 and subsequent cycles, participants received MK-8242 350 mg PO BID on Days 1-7 of each 21-day cycle.
  Interventions: Drug: MK-8242
- MK-8242 400 mg BID (Experimental): In Cycle 1, participants received MK-8242 400 mg administered PO BID on Days 1-6 and PO QD in the morning on Day 7 of the 21-day cycle to accommodate PK sampling. In Cycle 2 and subsequent cycles, participants received MK-8242 400 mg PO BID on Days 1-7 of each 21-day cycle.
  Interventions: Drug: MK-8242
- MK-8242 500 mg BID (Experimental): In Cycle 1, participants received MK-8242 500 mg administered PO BID on Days 1-6 and PO QD in the morning on Day 7 of the 21-day cycle to accommodate PK sampling. In Cycle 2 and subsequent cycles, participants received MK-8242 500 mg PO BID on Days 1-7 of each 21-day cycle.
  Interventions: Drug: MK-8242

INTERVENTIONS:
Drug: MK-8242 — 10 mg, 100 mg and 150 mg capsules
  Other Names: SCH 900242

SUMMARY:
This study is being done to evaluate the safety and pharmacokinetic profile of MK-8242 and its active metabolite (M16) in participants with advanced solid tumors. In Part 1 of the study, the study drug dose will be escalated to determine the maximum tolerated dose (MTD). In Part 2 of the study, the MTD will be confirmed and the recommended Phase 2 dose (RPTD) established; the effect of MK-8242 on liposarcoma and other tumor types will also be evaluated.

DETAILED DESCRIPTION:
Participants are considered to have completed the study after Cycle 12. Amendment 4 (14 April 2015) was done to allow participants on active treatment at the time the study was closed to enrollment to continue study treatment beyond Cycle 12 if deriving clinical benefit, at the Investigator's discretion.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed advanced solid tumor for which there are no effective standard therapy options
* Willing to provide tumor tissue for p53 wild type gene analysis
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
* Adequate organ function
* Female participants and male participants and their partners who are of childbearing potential must agree to abstain from sexual intercourse or to use an acceptable method of contraception during the study and for 90 days following the last dose of study drug
* At least one measurable lesion
* In Part 2, participants with liposarcoma must have a confirmed well-differentiated or de-differentiated histology

Exclusion criteria:

* Known treated or untreated leptomeningeal metastases, or metastatic central nervous system disease
* History of recent myocardial infarction (within the past year); or with unstable or uncontrolled angina, New York Heart Association (NYHA) Class III or IV congestive heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or clinically significant electrocardiogram (ECG) abnormality
* Uncontrolled active infection on optimal systemic treatment
* Clinically significant hepatitis or hepatitis C antibody positive, hepatitis B surface antigen positive, or human immunodeficiency virus (HIV) seropositive
* Persistent, unresolved common terminology criteria for adverse events (CTCAE v4.0) ≥Grade 2 drug-related toxicity associated with previous treatment except for alopecia
* Radiation therapy or other loco-regional therapy within 2 weeks prior to study
* Use of moderate and strong cytochrome P450 inhibitors or inducers within 1 week prior to study
* Chemotherapy or any investigational drug(s) within 4 weeks prior to study
* Known hypersensitivity to MK-8242 or its components
* Nursing, pregnant, or intention to become pregnant during the study
* Initiating bisphosphonate therapy or adjusting the bisphosphonate dose or regimen within 30 days of Cycle 1 Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-12-21 (Actual); Primary Completion 2014-09-15 (Actual); Study Completion 2015-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Wagner AJ, Banerji U, Mahipal A, Somaiah N, Hirsch H, Fancourt C, Johnson-Levonas AO, Lam R, Meister AK, Russo G, Knox CD, Rose S, Hong DS. Phase I Trial of the Human Double Minute 2 Inhibitor MK-8242 in Patients With Advanced Solid Tumors. J Clin Oncol. 2017 Apr 20;35(12):1304-1311. doi: 10.1200/JCO.2016.70.7117. Epub 2017 Feb 27. PMID 28240971

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MK-8242 60 mg BID | MK-8242 120 mg BID | MK-8242 170 mg BID | MK-8242 250 mg BID | MK-8242 300 mg BID | MK-8242 350 mg BID | MK-8242 400 mg BID | MK-8242 500 mg BID
Started | 1 | 6 | 3 | 7 | 3 | 6 | 16 | 6
Treated | 1 | 6 | 3 | 7 | 3 | 6 | 15 | 6
Completed | 1 | 4 | 2 | 3 | 2 | 3 | 6 | 2
Not Completed | 0 | 2 | 1 | 4 | 1 | 3 | 10 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 2 | 0 | 1 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 1 | 0 | 1 | 0 | 1 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0
Not completed — Not Treated | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- MK-8242 60 mg BID: In Cycle 1, participants received MK-8242 60 mg administered PO BID on Days 1-6 and PO QD in the morning on Day 7 of the 21-day cycle to accommodate PK sampling. In Cycle 2 and subsequent cycles, participants received MK-8242 60 mg PO BID on Days 1-7 of each 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | MK-8242 60 mg BID | MK-8242 120 mg BID | MK-8242 170 mg BID | MK-8242 250 mg BID | MK-8242 300 mg BID | MK-8242 350 mg BID | MK-8242 400 mg BID | MK-8242 500 mg BID | Total
Number analyzed (Participants) | 1 | 6 | 3 | 7 | 3 | 6 | 16 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.0 (NA) — Only 1 participant in population; no SD calculated. | 60.0 (11.0) | 68.3 (7.4) | 60.3 (11.4) | 53.3 (12.3) | 58.2 (10.2) | 63.9 (10.4) | 62.5 (12.8) | 61.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 3 | 1 | 2 | 6 | 3 | 19
  Male | 1 | 4 | 1 | 4 | 2 | 4 | 10 | 3 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as: any drug-related hematologic toxicity ≥ Grade 3 lasting ≥1 week, ≥ Grade 3 thrombocytopenia with bleeding, ≥ Grade 3 neutropenia with infection OR non-hematologic DLTs that were any Grade 3, 4, or 5 toxicity with the following exceptions/clarifications: 1) Grade 3 nausea, vomiting, diarrhea, and dehydration were excluded from the determination of DLT if, in the opinion of the investigator and sponsor, they occurred in a setting of inadequate treatment, 2) Grade 3 nausea, vomiting, diarrhea, and dehydration were each considered a DLT if they persisted despite 72 hours of maximal supportive care measures or 3) Any abnormal non-hematological laboratory value ≥ Grade 3 (that is not attributable to any other causes) was considered a DLT only if medical intervention was required to treat the participant, the abnormality led to hospitalization, or the abnormality persisted for ≥1 week.
Time Frame: Cycle 1 (21 days)
Population: The DLT-evaluable population consisted of participants who received at least one dose of MK-8242 and completed Cycle 1 of Part 1 (dose escalation) or the dose confirmation portion of Part 2, or discontinued due to toxicity.
Measure: Number; unit: Participants
Arm/Group | MK-8242 60 mg BID | MK-8242 120 mg BID | MK-8242 170 mg BID | MK-8242 250 mg BID | MK-8242 300 mg BID | MK-8242 350 mg BID | MK-8242 400 mg BID | MK-8242 500 mg BID
Number analyzed (Participants) | 1 | 6 | 3 | 7 | 3 | 6 | 15 | 6
Participants | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 4

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of MK-8242
Description: PK plasma samples were to be collected at the following time points: 0, 0.5, 1, 2, 4, 6, 8,and 12 hours after the first dose on Day 1; and 0, 0.5, 1, 2, 4, 6, 8, 12, 24 (Day 8) and 48 (Day 9) hours post-dose on Day 7.
Time Frame: Cycle 1, Day 1 pre-dose and through 24 hours post dose; Cycle 1 Day 7 pre-dose and through 48 hours post dose
Population: The All Participants as Treated (APaT) population consisted of all participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-8242 60 mg BID | MK-8242 120 mg BID | MK-8242 170 mg BID | MK-8242 250 mg BID | MK-8242 300 mg BID | MK-8242 350 mg BID | MK-8242 400 mg BID | MK-8242 500 mg BID
Number analyzed (Participants) | 1 | 5 | 3 | 6 | 3 | 6 | 14 | 6
nM
  Day 1 (n=1, 5, 3, 6, 3, 6, 14, 6) | 162 (NA) — Only 1 participant had PK parameter assessed; no geometric coefficient of variation was calculated. | 402 (101.2) | 813 (208.7) | 1210 (80.4) | 1320 (33.4) | 1510 (166.2) | 3820 (39.4) | 4240 (45.5)
  Day 7 (n=1, 5, 3, 6, 3, 5, 12, 3) | 150 (NA) — Only 1 participant had PK parameter assessed; no geometric coefficient of variation was calculated. | 551 (90.1) | 1680 (30.2) | 1030 (133.7) | 1720 (89.7) | 1930 (52.4) | 3070 (38.7) | 1800 (63.0)

3. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of MK-8242
Description: PK plasma samples were to be collected at the following time points: 0, 0.5, 1, 2, 4, 6, 8 and 12 hours after the first dose on Day 1; and 0, 0.5, 1, 2, 4, 6, 8, 12, 24 (Day 8) and 48 (Day 9) hours post-dose on Day 7.
Time Frame: Cycle 1, Day 1 pre-dose and through 12 hours postdose; Cycle 1 Day 7 pre-dose and through 48 hours post dose
Population: The APaT population consisted of all participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: Hours
Arm/Group | MK-8242 60 mg BID | MK-8242 120 mg BID | MK-8242 170 mg BID | MK-8242 250 mg BID | MK-8242 300 mg BID | MK-8242 350 mg BID | MK-8242 400 mg BID | MK-8242 500 mg BID
Number analyzed (Participants) | 1 | 5 | 3 | 6 | 3 | 6 | 14 | 6
Hours
  Day 1 (n=1, 5, 3, 6, 3, 6, 14, 6) | 2.03 [NA to NA] — Only 1 participant had PK parameter assessed; no full range was calculated. | 2.07 [1.95 to 6.08] | 4.30 [2.00 to 6.00] | 4.00 [2.00 to 4.27] | 2.18 [2.00 to 2.23] | 4.04 [2.00 to 4.08] | 2.00 [1.00 to 11.47] | 3.04 [2.00 to 8.00]
  Day 7 (n=1, 5, 3, 6, 3, 5, 12, 3) | 1.98 [NA to NA] — Only 1 participant had PK parameter assessed; no full range was calculated. | 4.00 [1.88 to 6.08] | 2.00 [2.00 to 4.00] | 3.23 [2.00 to 11.97] | 2.00 [2.00 to 2.00] | 4.00 [2.00 to 5.97] | 3.03 [2.00 to 6.92] | 2.08 [2.00 to 4.00]

4. Secondary Outcome: Area Under the Concentration Time Curve From Hour 0 to Hour 12 (AUC0-12) for MK-8242
Description: as for outcome 3
Time Frame: Cycle 1, Day 1 and Day 7, Hour 0 through Hour 12
Population: The APaT population consisted of all participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | MK-8242 60 mg BID | MK-8242 120 mg BID | MK-8242 170 mg BID | MK-8242 250 mg BID | MK-8242 300 mg BID | MK-8242 350 mg BID | MK-8242 400 mg BID | MK-8242 500 mg BID
Number analyzed (Participants) | 1 | 5 | 3 | 6 | 3 | 6 | 14 | 6
hr*nM
  Day 1 (n=1, 4, 1, 3, 3, 2, 12, 4) | 548 (NA) — Only 1 participant had PK parameter assessed; no geometric coefficient of variation was calculated. | 1820 (51.2) | 11000 (NA) — Only 1 participant had PK parameter assessed; no geometric coefficient of variation was calculated. | 5550 (100.1) | 5020 (45.4) | 6940 (110.7) | 16800 (45.3) | 24100 (46.0)
  Day 7 (n=1, 5, 3, 6, 3, 4, 12, 3) | 706 (NA) — Only 1 participant had PK parameter assessed; no geometric coefficient of variation was calculated. | 2450 (57.9) | 7190 (24.7) | 6710 (130.9) | 8720 (65.1) | 13100 (70.2) | 16500 (41.2) | 13400 (77.8)

5. Secondary Outcome: AUC at Time of Last Sample (AUClast) for MK-8242
Description: as for outcome 3
Time Frame: Cycle 1, Day 1 pre-dose and through 12 hours post dose; Cycle 1 Day 7 pre-dose and through 48 hours post dose
Population: The APaT population consisted of all participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | MK-8242 60 mg BID | MK-8242 120 mg BID | MK-8242 170 mg BID | MK-8242 250 mg BID | MK-8242 300 mg BID | MK-8242 350 mg BID | MK-8242 400 mg BID | MK-8242 500 mg BID
Number analyzed (Participants) | 1 | 5 | 3 | 6 | 3 | 6 | 14 | 6
hr*nM
  Day 1 (n=1, 5, 3, 6, 3, 6, 14, 6) | 509 (NA) — Only 1 participant had PK parameter assessed; no geometric coefficient of variation was calculated. | 1380 (72.0) | 3240 (131) | 5410 (69.0) | 4830 (49.7) | 6350 (152) | 16700 (41.9) | 17400 (84.7)
  Day 7 (n=1, 5, 3, 6, 3, 5, 12, 3) | 677 (NA) — Only 1 participant had PK parameter assessed; no geometric coefficient of variation was calculated. | 2260 (65.0) | 8290 (25.1) | 7590 (103) | 11300 (75.0) | 15100 (81.1) | 21400 (48.2) | 17300 (90.4)

ADVERSE EVENTS:
Time Frame: Up to approximately 10 months (Up to 30 days after last dose of study drug)
Description: The All Participants as Treated (APaT) population consisted of all participants who received at least one dose of study drug.
Arm/Group | MK-8242 60 mg BID | MK-8242 120 mg BID | MK-8242 170 mg BID | MK-8242 250 mg BID | MK-8242 300 mg BID | MK-8242 350 mg BID | MK-8242 400 mg BID | MK-8242 500 mg BID
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/6 | 0/3 | 2/7 | 1/3 | 3/6 | 5/15 | 4/6
Other Adverse Events (participants affected / at risk) | 1/1 | 6/6 | 3/3 | 7/7 | 3/3 | 6/6 | 15/15 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8242 60 mg BID (N=1) | MK-8242 120 mg BID (N=6) | MK-8242 170 mg BID (N=3) | MK-8242 250 mg BID (N=7) | MK-8242 300 mg BID (N=3) | MK-8242 350 mg BID (N=6) | MK-8242 400 mg BID (N=15) | MK-8242 500 mg BID (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8242 60 mg BID (N=1) | MK-8242 120 mg BID (N=6) | MK-8242 170 mg BID (N=3) | MK-8242 250 mg BID (N=7) | MK-8242 300 mg BID (N=3) | MK-8242 350 mg BID (N=6) | MK-8242 400 mg BID (N=15) | MK-8242 500 mg BID (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 10 (22) | 3 (4)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (6) | 0 (0) | 2 (7) | 9 (23) | 2 (6)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presbyopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coeliac artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (4) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (3) | 3 (3) | 2 (4) | 3 (4) | 13 (23) | 5 (15)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (10) | 3 (10) | 5 (11) | 3 (10) | 5 (15) | 12 (21) | 5 (11)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (4) | 4 (10) | 1 (2) | 4 (7) | 7 (11) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 4 (7) | 3 (6) | 6 (7) | 2 (5) | 4 (10) | 12 (17) | 6 (14)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal bacterial overgrowth (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coagulation time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (7)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 1 (1) | 5 (6) | 1 (2) | 3 (6) | 11 (17) | 3 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (7) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allodynia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (6) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.